CLINICAL TRIAL: NCT00193544
Title: Phase II Trial of Arsenic Trioxide and Thalidomide in the Treatment of Patients With Refractory Multiple Myeloma
Brief Title: Arsenic Trioxide and Thalidomide in the Treatment of Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: CTI BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 03
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Arsenic Trioxide; Thalidomide

INTERVENTIONS:
Drug: Arsenic Trioxide
Drug: Thalidomide

SUMMARY:
In this trial, we plan to evaluate further the role of arsenic trioxide in the treatment of patients with refractory multiple myeloma. Arsenic trioxide will be used in combination with thalidomide. Although both drugs have a similar mechanism of action, it is likely that the mechanisms may be additive or synergistic. Since neither drug produces much myelosuppression, this combination regimen should be tolerable in patients with compromised marrow function due to involvement with myeloma and/or previous cytotoxic chemotherapy

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Arsenic Trioxide + Thalidomide

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Confirmed diagnosis of multiple Myeloma
* Received at least one previous chemotherapy regimen at most 3 previous
* Thalidomide with or without dexamethasone without chemotherapy will not factor in to total number of regimens.
* Age at least 18 years years
* Able to perform activities of daily living with minimal assistance
* Life expectancy more than 3 months
* Adequate bone marrow, liver and kidney function
* Must give written informed consent in order to participate.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Women pregnant or lactating.
* Pre-existing moderate neuropathy
* Patients with significant underlying cardiac dysfunction
* Uncontrolled hypercalcemia
* Active serious infections not controlled by antibiotics
* History of grand mal seizures (other than infantile febrile seizures)
* Receiving other medications that prolong the QT interval.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-03; Primary Completion 2005-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Overall survival
Time to progression
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC